CLINICAL TRIAL: NCT02309944
Title: Negative Pressure Wound Therapy in Obese Gynecologic Oncology Patients: A Randomized Controlled Trial
Brief Title: Negative Pressure Wound Therapy in Obese Gynecologic Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013NTLS073
Record Dates: First submitted 2014-11-19; First posted 2014-12-05 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Complications; Obesity; Gynecologic Neoplasms
Keywords: Wound Healing; Obesity; Gynecologic Surgery; Gynecologic Neoplasms; Surgical Complications
MeSH Terms: conditions — Postoperative Complications; Obesity; Genital Neoplasms, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Wound Closure (Active Comparator): Standard surgical closure of the fascia and skin.
  Interventions: Procedure: Standard Wound Closure
- Negative Pressure Wound Therapy (Experimental): Standard surgical closure as used by the standard of care group plus placement of the Prevena™ Incision Management System over the closed incision.
  Interventions: Procedure: Standard Wound Closure; Device: Prevena™ Incision Management System

INTERVENTIONS:
Procedure: Standard Wound Closure — The standard surgical closure consists of closure of the fascia with a looped polydioxanone (PDS) suture in a running fashion either in with the use of a mass closure technique or a Smead Jones closure at the discretion of the operating surgeon, closure of the subcutaneous space if >2 cm deep, followed by staple or suture closure of the skin.
Device: Prevena™ Incision Management System — At the close of surgery, the Prevena™ Incision Management System will be placed over the closed incision. It will be removed on post-operative day 2 or 3 as clinically indicated and prior to the patient's discharge from the hospital.
  Arms: Negative Pressure Wound Therapy

SUMMARY:
The purpose of the study is to test whether the use of a new wound closure technique can decrease the rates of wound complications in obese cancer patients.

DETAILED DESCRIPTION:
Most gynecologic and many intra-abdominal malignancies are treated with an initial surgical procedure. There has been a dramatic increase in obesity rates in the US with more than one third of US adults being obese (Body Mass Index (BMI) of > 30kg/m2). There is a direct link between obesity and wound complications following surgery with an increasing BMI leading to increasing rates of complications. Negative pressure wound therapy (NPWT) is a system that utilizes sub-atmospheric pressure to improve wound healing by increasing the formation of granulation tissue. NPWT has been shown to improve outcomes in both the orthopedic and cardiothoracic surgery populations. To date, there is no prospective study evaluating the application of prophylactic NPWT in laparotomy patients.

This study will be a randomized clinical trial. Patients will be enrolled at the time of consent for laparotomy for suspected gynecologic malignancy. Participants will be randomized to one of two groups: 1) Standard closure group (control arm): closure of the fascia, subcutaneous tissue and skin per the surgeon's standard method; or 2) NPWT group (study arm): closure of the fascia, subcutaneous tissue and skin per the surgeon's standard method + placement of a negative pressure wound therapy device over the closed incision for 2-3 days, with removal of the device prior to hospital discharge. The rate of wound complications for two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected gynecologic or other abdominal malignancy (such as colorectal, liver, pancreatic, kidney and stomach) for which laparotomy is planned
* Obese - defined as a Body Mass Index (BMI) ≥ 35 kg/m2 as calculated in the Epic computer record

Exclusion Criteria:

* Known true tape allergy
* Sensitivity to silver
* History of intolerance to Negative Pressure Wound Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna G. Teoh, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 participants originally consented, one withdrew consent and 11 did not return updated HIPAA forms and therefore could not be included in the analysis
Period: Overall Study
Arm/Group | Standard Wound Closure | Negative Pressure Wound Therapy
Started | 38 | 43
Completed | 38 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Wound Closure | Negative Pressure Wound Therapy | Total
Number analyzed (Participants) | 38 | 43 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.9) | 59.6 (11.4) | 59.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 36 | 41 | 77
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 34 | 32 | 66
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 38 | 43 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Wound Complications (Wound Dehiscence or Infection)
Time Frame: one month after surgery
Population: Follow up data is not available for 2 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Wound Closure | Negative Pressure Wound Therapy
Number analyzed (Participants) | 37 | 42
Participants
  No | 25 | 33
  Yes | 12 | 9
Statistical Analysis 1: Comparison: Standard Wound Closure vs Negative Pressure Wound Therapy; Negative Pressure Wound Therapy vs. Standard Wound Closure; Test type: Superiority; p = 0.27, Chi-squared
Statistical Analysis 2: Comparison: Standard Wound Closure vs Negative Pressure Wound Therapy; Negative Pressure Wound Therapy vs. Standard Wound Closure; Test type: Superiority; p = 0.24, Regression, Logistic; Multivariate Model (adjusted for ascites and previous laparotomy)

2. Secondary Outcome: Time From Surgery to Starting Adjuvant Therapy Among Those With Confirmed Malignancies
Time Frame: up to 20 weeks
Population: Only those participants who received adjuvant therapies were analyzed in both arms. Rest of the patients didn't have cancer that required subsequent therapies.
Measure: Median (Full Range); unit: days
Arm/Group | Standard Wound Closure | Negative Pressure Wound Therapy
Number analyzed (Participants) | 19 | 17
days | 37 [13 to 132] | 28 [13 to 90]

ADVERSE EVENTS:
Time Frame: Upto 12 weeks after surgery
Arm/Group | Standard Wound Closure | Negative Pressure Wound Therapy
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/43
Serious Adverse Events (participants affected / at risk) | 7/38 | 17/43
Other Adverse Events (participants affected / at risk) | 5/38 | 3/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Wound Closure (N=38) | Negative Pressure Wound Therapy (N=43)
postop ileus (Gastrointestinal disorders) | 3 | 6
pulmonary embolism (Blood and lymphatic system disorders) | 0 | 2
Anastomotic leak (Gastrointestinal disorders) | 0 | 1
Vaginal cuff dehiscence (Skin and subcutaneous tissue disorders) | 0 | 1
atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 | 0
Postop hypotension (Cardiac disorders) | 1 | 2
Pelvic abscess (Infections and infestations) | 1 | 0
malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Superficial wound infection, requiring readmission (Infections and infestations) | 0 | 2
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowel perforation (Gastrointestinal disorders) | 1 | 0
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Wound Closure (N=38) | Negative Pressure Wound Therapy (N=43)
Hospital-acquired pneumonia (Infections and infestations) | 1 | 0
Postop hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Genital yeast infection (Infections and infestations) | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 1
acute kidney injury (Renal and urinary disorders) | 0 | 1
Superficial wound infection (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02309944/Prot_SAP_000.pdf